CLINICAL TRIAL: NCT04886180
Title: Evaluation of Oxiris Membrane as a Treatment for Ischemia-reperfusion Syndrome in Cardiogenic Shock Treated With Extracorporeal Life Support (ECMO/ECLS): A Randomized Pilot Study ECMORIX
Acronym: ECMORIX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NGUYEN 2020-2
Record Dates: First submitted 2021-05-10; First posted 2021-05-13 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Cardiogenic Shock
MeSH Terms: conditions — Shock, Cardiogenic | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental)
  Interventions: Device: Oxiris membrane; Biological: Blood tests
- Control (Active Comparator)
  Interventions: Device: Prismaflex membrane; Biological: Blood tests

INTERVENTIONS:
Device: Oxiris membrane — Hemofiltration treatment with Oxiris membrane connected to the ECLS circuit for 24 hours.
  Arms: Experimental
Device: Prismaflex membrane — Treatment by hemofiltration with PrismaFlex ST150 membrane connected to the ECLS circuit for 24 hours.
  Arms: Control
Biological: Blood tests — Blood tests before and just after membrane placement and at H6, H24, H48 and H72 after membrane placement

SUMMARY:
The Oxiris membrane is an AN-69 membrane whose surface is treated with polyethyleneimine (PEI) grafted with heparin. This property allows the removal of lipopolysaccharide and cytokines from the blood. During septic shock, this membrane has shown its effectiveness and made it possible to decrease the doses of vasopressors administered, thus limiting the negative consequences of their use (low mesenteric flow in particular). Moreover, the literature suggests that the use of the Oxiris membrane does not lead to side effects or specific and serious complications, in comparison with conventional extra-renal purification membranes. To our knowledge (Pubmed, clinicaltrial) there are no data in patients in cardiogenic shock assisted by ECLS.

The research hypothesis is that the early addition of an Oxiris membrane to the ECLS circuit allows the removal of lipopolysaccharides and pro-inflammatory cytokines, thus controlling the inflammatory cascade and limiting vasoplegia and organ failure.

ELIGIBILITY:
Inclusion Criteria:

* Trusted person or relative who has given oral consent or emergency consent
* Person of legal age
* Patient receiving ECLS for refractory cardiogenic shock requiring continuous renal replacement therapy
* Included within 12 hours of ECLS initiation

Exclusion Criteria:

* Person not affiliated to national health insurance
* Person under legal protection (curatorship, guardianship)
* Person under court order
* Pregnant or breastfeeding woman
* Minor
* Severe hemorrhage under ECLS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2023-03-10 (Actual); Study Completion 2023-03-10 (Actual)

PRIMARY OUTCOMES:
Plasma concentration of lipopolysaccharides | 24 hours after addition of the membrane

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France

REFERENCES:
- [Derived] Nguyen M, Alvarez M, Evezard C, Berthoud V, Leleu D, Pais-De-Barros JP, Bouchot O, Abou-Arab O, Bouhemad B, Masson D, Gautier T, Guinot PG. Endotoxin removal by the OXIRIS filter for cardiogenic shock requiring veno-arterial extra-corporeal life support: the ECMORIX randomized controlled trial. Ann Intensive Care. 2025 Jul 8;15(1):92. doi: 10.1186/s13613-025-01499-z. PMID 40627256
- [Derived] Andrei S, Nguyen M, Berthoud V, Morgant MC, Bouhemad B, Guinot PG; ECMORIX Study Group. Evaluation of the Oxiris Membrane in Cardiogenic Shock Requiring Extracorporeal Membrane Oxygenation Support: Study Protocol for a Single Center, Single-Blind, Randomized Controlled Trial. Front Cardiovasc Med. 2021 Oct 11;8:738496. doi: 10.3389/fcvm.2021.738496. eCollection 2021. PMID 34708091